CLINICAL TRIAL: NCT01847326
Title: Nab-Paclitaxel-based Re-induction Chemotherapy Followed by Response-stratified Chemoradiotherapy in Patients With Previously Treated Squamous Cell Carcinoma of the Head and Neck.
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation and Carboplatin Followed By Chemoradiation in Treating Patients With Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1554; NCI-2012-02179 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-04-19; First posted 2013-05-06 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Tongue Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Carboplatin; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Fluorouracil; Hydroxyurea; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (induction therapy and AFHX or AXX) (Experimental): See Detailed Description
  Interventions: Drug: carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: fluorouracil; Drug: hydroxyurea; Procedure: therapeutic conventional surgery; Radiation: radiation therapy; Radiation: hyperfractionated radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: hydroxyurea — Given PO
  Other Names: HU; HYD; Hydrea; Hydroxycarbamide; Hydurea
Procedure: therapeutic conventional surgery — Undergo surgical resection
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Radiation: hyperfractionated radiation therapy — Undergo hyperfractionated radiation therapy
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of paclitaxel albumin-stabilized nanoparticle formulation when given together with carboplatin followed by chemoradiation in treating patients with recurrent head and neck cancer. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, carboplatin, fluorouracil, and hydroxyurea, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving paclitaxel albumin-stabilized nanoparticle formulation followed by chemoradiation therapy may be an effective treatment for head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) when given in combination with FHX (5 fluorouracil [fluorouracil], hydroxyurea and twice daily radiation, in good induction responders) and of nab-paclitaxel added to hypofractionated radiotherapy for poor responders.

II. To explore the feasibility of a more rapid palliative chemoradiotherapy approach inpatients with refractory disease as demonstrated by failure to respond to initial chemotherapy.

III. To explore the role of induction chemotherapy as a predictive tool for definitive head and neck cancer management of previously treated patients.

SECONDARY OBJECTIVES:

I. Progression-free survival (PFS) (time to disease progression or death from any cause) on both study arms.

II. Overall survival and response rates in both arms.

TERTIARY OBJECTIVES:

I. To determine the correlation of secreted protein, acidic, cysteine-rich (SPARC) expression in head and neck cancer and response to therapy.

OUTLINE: This is a dose-escalation study of paclitaxel albumin-stabilized nanoparticle formulation.

RE-INDUCTION THERAPY (WEEKS 1-6): Patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 1. Courses repeat every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving good response undergo surgical resection and proceed to chemoradiation within 4-6 weeks.

AFHX REGIMEN: Patients achieving response to re-induction therapy receive hydroxyurea orally (PO) every 12 hours for 6 days (11 doses) beginning on day 0, fluorouracil IV continuously over 120 hours beginning on day 0, and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1. Patients also undergo radiation therapy twice daily (BID) on days 1-5. Courses repeat every 14 days for 5 weeks in the absence of disease progression or unacceptable toxicity.

PACLITAXEL + RADIATION (AXX) REGIMEN: Patients not achieving response to re-induction therapy receive paclitaxel albumin-stabilized nanoparticle formulation IV and undergo hypofractionated radiation therapy on day 1. Courses repeat every 7 days for 5 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 3 months, every 3 months for 2 years, every 6 months for 2 years, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of recurrent head and neck cancer requiring regional therapy
* Recurrent or second primary, previously irradiated squamous cell carcinoma of the head and neck (SCCHN) without clinically measurably metastatic disease
* Prior radiation therapy completed >= 4 months, and/or chemotherapy completed >= 1 month before study entry, and patient should have recovered from any adverse effects
* Predominance of disease that is amenable to radiotherapy
* Measurable disease prior to induction chemotherapy
* Eastern Cooperative Oncology Group performance status of one or less
* Life expectancy of greater than 12 weeks
* Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment
* Negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test at screening for patients of childbearing potential
* Patients must have < grade 2 pre-existing peripheral neuropathy (per Common Terminology Criteria for Adverse Events [CTCAE])
* Leukocyte >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 1000,000/ul
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x institutional upper limit of normal
* Creatinine clearance (CrCl) > 45 mL/min

Exclusion Criteria:

* Previously untreated patients with locoregional-only disease are not eligible
* Patients who have had chemotherapy within 4 weeks prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical composition agents used in the study
* Patients with pre-existing grade 2 or greater peripheral neuropathy, defined as sensory alteration or paresthesia (including tingling), interfering with function
* Uncontrolled intercurrent illness including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of paclitaxel albumin-stabilized nanoparticle formulation in combination with fluorouracil, hydroxyurea, and radiation therapy, determined according to incidence of DLT graded using the National Cancer Institute (NCI) CTCAE 4.0 | 4 weeks
Recommended phase II dose of paclitaxel albumin-stabilized nanoparticle formulation in combination with radiation therapy, determined according to incidence of DLT graded using the NCI CTCAE 4.0 | 4 weeks

SECONDARY OUTCOMES:
PFS | The time from the date of registration to the date of progressive disease or death, assessed up to 1 year
  Statistical significance will be determined by a two-sided P value =< 0.05. Progression-free survival curves will be calculated using the Kaplan-Meier method, and median progression-free survival time, along with 90% confidence intervals will be derived using the procedure described in Brookmeyer and Crowley.
Overall survival | The time from the date of registration to the date of death, assessed up to 1 year
  Statistical significance will be determined by a two-sided P value =< 0.05. Overall survival curves will be calculated using the Kaplan-Meier method, and median overall survival time, along with 90% confidence intervals will be derived using the procedure described in Brookmeyer and Crowley.
Objective response rate (complete response [CR] + partial response [PR]) | Up to 1 year
  The objective response rate (CR + PR) and associated 90% confidence interval will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas de Souza, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Rosenberg AJ, Agrawal N, Pearson AT, Gooi Z, Blair E, Portugal L, Cursio JF, Juloori A, Chin J, Rouse K, Villaflor VM, Seiwert TY, Izumchenko E, Lingen MW, Haraf DJ, Vokes EE. Phase I study of nab-paclitaxel-based induction followed by nab-paclitaxel-based concurrent chemotherapy and re-irradiation in previously treated head and neck squamous cell carcinoma. Br J Cancer. 2022 Nov;127(8):1497-1506. doi: 10.1038/s41416-022-01941-0. Epub 2022 Aug 9. PMID 35945244